CLINICAL TRIAL: NCT00422097
Title: A Phase I Study of Ixabepilone Administered as a Daily Oral Dose on 5 Successive Days Every 21 Days in Subjects With Advanced Cancer
Brief Title: A Phase I Study of Oral Ixabepilone in Subjects With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: R-Pharm (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CA163-111
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Results first posted 2011-04-20 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — ixabepilone; Famotidine; Food

ARMS (8):
- Ixabepilone, 5 mg/d (Experimental): If none of first 3 participants experiences a dose-limiting toxicity (DLT) during the first 21-day cycle, a new cohort is opened at the next dose level (5-mg increments). If 2 or more of the first 3 participants experience a DLT within the first 21-day course, the dose level will be considered above the maximum tolerated dose (MTD). If 1 of the first 3 participants experiences a DLT, an additional 3 participants will be enrolled at this dose level for a total of 6 participants. If 2 or more of the 6 participants (or 1/3 or more of a cohort with more than 6 participants) experience a DLT, this dose level will be considered above the MTD.
  Interventions: Drug: Ixabepilone, 5 mg/d
- Ixabepilone, 10 mg/d (Experimental): If none of first 3 participants experiences a DLT during the first 21-day cycle, a new cohort is opened at the next dose level (5-mg increments). If 2 or more of the first 3 participants experience a DLT within the first 21-day course, the dose level will be considered above the MTD. If 1 of the first 3 participants experiences a DLT, an additional 3 participants will be enrolled at this dose level for a total of 6 participants. If 2 or more of the 6 participants (or 1/3 or more of a cohort with more than 6 participants) experience a DLT, this dose level will be considered above the MTD.
  Interventions: Drug: Ixabepilone, 10 mg/d
- Ixabepilone, 15 mg/d (Experimental): If none of first 3 participants experiences a DLT during the first 21-day cycle, a new cohort is opened at the next dose level (5-mg increments). If 2 or more of the first 3 participants experience a DLT within the first 21-day course, the dose level will be considered above the MTD. If 1 of the first 3 participants experiences a DLT, an additional 3 participants will be enrolled at this dose level for a total of 6 participants. If 2 or more of the 6 participants (or 1/3 or more of a cohort with more than 6 participants) experience a DLT, this dose level will be considered above the MTD.
  Interventions: Drug: Ixabepilone, 15 mg/d
- Ixabepilone, 20 mg/d (Experimental): If none of first 3 participants experiences a DLT during the first 21-day cycle, a new cohort is opened at the next dose level (5-mg increments). If 2 or more of the first 3 participants experience a DLT within the first 21-day course, the dose level will be considered above the MTD. If 1 of the first 3 participants experiences a DLT, an additional 3 participants will be enrolled at this dose level for a total of 6 participants. If 2 or more of the 6 participants (or 1/3 or more of a cohort with more than 6 participants) experience a DLT, this dose level will be considered above the MTD.
  Interventions: Drug: Ixabepilone, 20 mg/d
- Ixabepilone, 25 mg/d (Experimental): If none of first 3 participants experiences a DLT during the first 21-day cycle, a new cohort is opened at the next dose level (5-mg increments). If 2 or more of the first 3 participants experience a DLT within the first 21-day course, the dose level will be considered above the MTD. If 1 of the first 3 participants experiences a DLT, an additional 3 participants will be enrolled at this dose level for a total of 6 participants. If 2 or more of the 6 participants (or 1/3 or more of a cohort with more than 6 participants) experience a DLT, this dose level will be considered above the MTD.
  Interventions: Drug: Ixabepilone, 25 mg/d
- Ixabepilone, 30 mg/d (Experimental): If none of first 3 participants experiences a DLT during the first 21-day cycle, a new cohort is opened at the next dose level (5-mg increments). If 2 or more of the first 3 participants experience a DLT within the first 21-day course, the dose level will be considered above the MTD. If 1 of the first 3 participants experiences a DLT, an additional 3 participants will be enrolled at this dose level for a total of 6 participants. If 2 or more of the 6 participants (or 1/3 or more of a cohort with more than 6 participants) experience a DLT, this dose level will be considered above the MTD.
  Interventions: Drug: Ixabepilone, 30 mg/d
- Ixabepilone, 25 mg, with famotidine (Experimental): Following identification of MTD, participants who completed Cycle 1 and treated at the ixabepilone MTD (25 mg/d) will crossover to Cycle 2 in which they receive famotidine, 40 mg on Day 1.
  Interventions: Drug: Ixabepilone, 25 mg, with famotidine
- Ixabepilone, 25 mg, with food (Experimental): Following identification of MTD, participants who completed Cycle 1 and treated at the ixabepilone MTD (25 mg/d) will crossover to Cycle 2 in which they receive a low-fat meal on Day 1.
  Interventions: Drug: Ixabepilone, 25 mg, with food

INTERVENTIONS:
Drug: Ixabepilone, 5 mg/d — Ixabepilone, 5 mg, administered orally once daily on Days 1 through 5 every 21 days. Dose increased by 5 mg for each subsequent treatment group until disease progression, unacceptable toxicity, or participant refusal. No dose escalation within each treatment group. On all dosing days in Cycle 1, participants must fast at least 4 hours before and 4 hours after treatment.
  Arms: Ixabepilone, 5 mg/d
Drug: Ixabepilone, 10 mg/d — Ixabepilone, 10 mg, administered orally once daily on Days 1 through 5 every 21 days. Dose increased by 5 mg for each subsequent treatment group until disease progression, unacceptable toxicity, or participant refusal. No dose escalation within each treatment group. On all dosing days in Cycle 1, participants must fast at least 4 hours before and 4 hours after treatment.
  Arms: Ixabepilone, 10 mg/d
Drug: Ixabepilone, 15 mg/d — Ixabepilone, 15 mg, administered orally once daily on Days 1 through 5 every 21 days. Dose increased by 5 mg for each subsequent treatment group until disease progression, unacceptable toxicity, or participant refusal. No dose escalation within each treatment group. On all dosing days in Cycle 1, participants must fast at least 4 hours before and 4 hours after treatment.
  Arms: Ixabepilone, 15 mg/d
Drug: Ixabepilone, 20 mg/d — Ixabepilone, 20 mg, administered orally once daily on Days 1 through 5 every 21 days. Dose increased by 5 mg for each subsequent treatment group until disease progression, unacceptable toxicity, or participant refusal. No dose escalation within each treatment group. On all dosing days in Cycle 1, participants must fast at least 4 hours before and 4 hours after treatment.
  Arms: Ixabepilone, 20 mg/d
Drug: Ixabepilone, 25 mg/d — Ixabepilone, 25 mg, administered orally once daily on Days 1 through 5 every 21 days. Dose increased by 5 mg for each subsequent treatment group until disease progression, unacceptable toxicity, or participant refusal. No dose escalation within each treatment group. On all dosing days in Cycle 1, participants must fast at least 4 hours before and 4 hours after treatment.
  Arms: Ixabepilone, 25 mg/d
Drug: Ixabepilone, 30 mg/d — Ixabepilone, 30 mg, administered orally once daily on Days 1 through 5 every 21 days. Dose increased by 5 mg for each subsequent treatment group until disease progression, unacceptable toxicity, or participant refusal. No dose escalation within each treatment group. On all dosing days in Cycle 1, participants must fast at least 4 hours before and 4 hours after treatment.
  Arms: Ixabepilone, 30 mg/d
Drug: Ixabepilone, 25 mg, with famotidine — Participants crossed over from Cycle 1 to receive famotidine, 40 mg, in an oral dose given 2 hours before ixabepilone, 25 mg, on Day 1 of Cycle 2 only.
  Arms: Ixabepilone, 25 mg, with famotidine
Drug: Ixabepilone, 25 mg, with food — Participants consume a low-fat meal starting 30 minutes before dose administration on Day 1 of Cycle 2. Food consumed within 30 minutes. Administration of the total oral dose should not exceed more than 10 minutes from start to finish.
  Arms: Ixabepilone, 25 mg, with food

SUMMARY:
This study will determine the maximum tolerated dose of oral ixabepilone administered for 5 successive days every 21 days in participants with advanced cancer. The safety, tolerability, and pharmacokinetics of ixabepilone in the body will be studied. In addition, this study will assess preliminary evidence of the effect of food and famotidine on the pharmacokinetics of oral ixabepilone.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of solid tumor malignancy unresponsive to current treatment options
* Measurable or nonmeasurable disease as defined by Response Evaluation Criteria in Solid Tumors
* Lapse of at least 1 week since minor surgery and of at least 3 weeks since major surgery and radiation therapy
* Eastern Cooperative Oncology Group performance status of 0-1
* Lapse of at least 4 weeks since immunotherapy or chemotherapy
* Negative pregnancy test result within 72 hours of study drug administration for any woman of childbearing potential (WOCBP)

Exclusion Criteria:

* WOCBP unable or unwilling to use birth control during study and for up to 4 weeks after study completion
* Women who are pregnant or breastfeeding
* Fertile men not using effective birth control with partners who are WOCBP
* Gastrointestinal(GI) disease or GI tract surgery that could impact drug absorption
* Inability to swallow capsules
* Inability to be venipunctured or to tolerate venous access
* Known symptomatic brain metastases
* Common Terminology Criteria for Adverse Events Grade 2 or greater neuropathy or history of Grade 3 or greater neuropathy
* Psychiatric conditions inhibiting compliance with protocol requirements
* Uncontrolled medical disorder or active infection that would impair participant's ability to receive protocol therapy or whose control may be jeopardized by the study treatment protocol
* Inadequate hematologic, hepatic, or renal function
* History of significant drug allergy
* Previous exposure to ixabepilone
* Exposure to any investigational drug or placebo within 4 weeks of enrollment
* Concurrent chemotherapy regimen
* Use of cytochrome P4503A4 inhibitors or inducers within 2 weeks of treatment initiation (unless approved by medical monitor)
* Use of steroids (except as antiemetic)
* Prisoners or subjects involuntarily detained for treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-01; Primary Completion 2009-08 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Georgetown University Medical Center Lombardi Cancer Center, Washington D.C., District of Columbia
  - Wayne State University (Hwcrc), Detroit, Michigan

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 58 enrolled, 44 received treatment: 10 no longer met enrollment criteria (2 brain metastases, 2 bowel obstruction, 1 high aspartame aminotransferase [AST], 1 high AST/alanine transaminase, 2 low platelets, 1 hospitalized, 1 gastric adverse event [AE]); 2 withdrew consent/changed mind; 1 AE; 1 sponsor administrative reason.
Groups:
- Ixabepilone, 5 mg/d: Ixabepilone, 5 mg, given once daily in an oral dose on Days 1 through 5 every 21 days. If none of the first 3 participants experiences a dose-limiting toxicity (DLT) in the first 21-day course, a new cohort is opened at the next dose level (10 mg/d). On all dosing days in Cycle 1, participants must fast at least 4 hours before and 4 hours after treatment. For Cycles 2 and greater, participants must fast 1 hour before and 2 hours after the dose.
- Ixabepilone, 10 mg/d: Ixabepilone, 10 mg, given once daily in an oral dose on Days 1 through 5 every 21 days. If none of the first 3 participants experiences a DLT during the first 21-day course, a new cohort is opened at the next dose level (15 mg/d). If 1 of the first 3 participants experiences a DLT, an additional 3 participants will be enrolled at this dose level for a total of 6 participants. On all dosing days in Cycle 1, participants must fast at least 4 hours before and 4 hours after treatment. For Cycles 2 and greater, participants must fast 1 hour before and 2 hours after the dose.
- Ixabepilone, 15 mg/d: Ixabepilone, 15 mg, given once daily in an oral dose on Days 1 through 5 every 21 days. If none of the first 3 participants experiences a DLT during the first 21-day course, a new cohort is opened at the next dose level (20 mg/d). If 1 of the first 3 participants experiences a DLT, an additional 3 participants will be enrolled at this dose level for a total of 6 participants. On all dosing days in Cycle 1, participants must fast at least 4 hours before and 4 hours after treatment. For Cycles 2 and greater, participants must fast 1 hour before and 2 hours after the dose.
- Ixabepilone, 20 mg/d: Ixabepilone, 20 mg, given daily in oral doses on Days 1 through 5 every 21 days. If none of the first 3 participants experiences a DLT during the first 21-day course, a new cohort is opened at the next dose level (25 mg/d). On all dosing days in Cycle 1, participants must fast at least 4 hours before and 4 hours after treatment. For Cycles 2 and greater, participants must fast 1 hour before and 2 hours after the dose.
- Ixabepilone, 25 mg/d: Ixabepilone, 25 mg/d, given once daily in an oral dose on Days 1 through 5 every 21 days. If none of the first 3 participants experiences a DLT in the first 21-day course, a new cohort is opened at the next dose level (30 mg/d). If 1 of the first 3 participants experiences a DLT, an additional 3 participants will be enrolled at this dose level for a total of 6 participants. If 2 or more of the 6 participants (or 1/3 or more of a cohort with more than 6 participants) experience a DLT, this dose level will be considered above the MTD. The MTD is the maximum dose that can be given to 6 participants without producing a DLT in more than 1 participant (or fewer than 1/3 if the cohort has more than 6 participants). More participants may be enrolled at any level to provide additional safety data. On all dosing days in Cycle 1, participants must fast at least 4 hours before and 4 hours after treatment. For Cycles 2 and greater, participants must fast 1 hour before and 2 hours after the dose.
- Ixabepilone, 30 mg/d: Ixabepilone, 30 mg, given daily orally on Days 1 through 5 every 21 days. If 2 or more of the first 3 participants experience a DLT within the first 21-day course, this dose level will be considered above the MTD. If 1 of the first 3 participants experiences a DLT, an additional 3 participants will be enrolled at this dose level for a total of 6 participants. If 2 or more of the 6 participants (or 1/3 or more of a cohort with more than 6 participants) experience a DLT, this dose level will be considered above the MTD (the maximum dose that can be given to 6 participants without producing a DLT in more than 1 [or fewer than 1/3 if more than 6 participants in cohort)]. On all dosing days in Cycle 1, participants to fast at least 4 hours before and 4 hours after treatment. For Cycles 2 and greater, participants must fast 1 hour before and 2 hours after the dose.
- Ixabepilone, MTD (25 mg), With Famotidine: Cohort opened for Cycle 2, once ixabepilone MTD (25 mg) determined. In Cycle 1, participants received ixabepilone, 25 mg, alone, orally once per day on Days 1 through 21. Then participants crossed over to receive famotidine wirh ixabepilone in Cycle 2. Prior to dosing on Day 1 of Cycle 2, famotidine, 40 mg, administered in an oral dose 2 hours before ixabepilone 25-mg dose.
- Ixabepilone, MTD (25 mg), With Food: Cohort opened for Cycle 2, after ixabepilone MTD (25 mg) determined. In Cycle 1, participants received ixabepilone, 25 mg, once daily in an oral dose on Days 1 through 5. On all dosing days in Cycle 1, participants fasted at least 4 hours before and 4 hours after dosing. Then participants crossed over to Cycle 2. On Day 1 of Cycle 2, participants allowed a low-fat meal. Participants ingest the specified meal within a 30-minute period and receive ixabepilone, 25 mg, 30 minutes after start of the meal. For the duration of Cycle 2, participants fast 1 hour before and 2 hours after ixabepilone dose.
Period: Dose Level 1
Arm/Group | Ixabepilone, 5 mg/d | Ixabepilone, 10 mg/d | Ixabepilone, 15 mg/d | Ixabepilone, 20 mg/d | Ixabepilone, 25 mg/d | Ixabepilone, 30 mg/d | Ixabepilone, MTD (25 mg), With Famotidine | Ixabepilone, MTD (25 mg), With Food
Started | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Level 2
Arm/Group | Ixabepilone, 5 mg/d | Ixabepilone, 10 mg/d | Ixabepilone, 15 mg/d | Ixabepilone, 20 mg/d | Ixabepilone, 25 mg/d | Ixabepilone, 30 mg/d | Ixabepilone, MTD (25 mg), With Famotidine | Ixabepilone, MTD (25 mg), With Food
Started | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Still on treatment | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Level 3
Arm/Group | Ixabepilone, 5 mg/d | Ixabepilone, 10 mg/d | Ixabepilone, 15 mg/d | Ixabepilone, 20 mg/d | Ixabepilone, 25 mg/d | Ixabepilone, 30 mg/d | Ixabepilone, MTD (25 mg), With Famotidine | Ixabepilone, MTD (25 mg), With Food
Started | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Level 4
Arm/Group | Ixabepilone, 5 mg/d | Ixabepilone, 10 mg/d | Ixabepilone, 15 mg/d | Ixabepilone, 20 mg/d | Ixabepilone, 25 mg/d | Ixabepilone, 30 mg/d | Ixabepilone, MTD (25 mg), With Famotidine | Ixabepilone, MTD (25 mg), With Food
Started | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Level 5
Arm/Group | Ixabepilone, 5 mg/d | Ixabepilone, 10 mg/d | Ixabepilone, 15 mg/d | Ixabepilone, 20 mg/d | Ixabepilone, 25 mg/d | Ixabepilone, 30 mg/d | Ixabepilone, MTD (25 mg), With Famotidine | Ixabepilone, MTD (25 mg), With Food
Started | 0 | 0 | 0 | 0 | 23 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 23 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Level 6
Arm/Group | Ixabepilone, 5 mg/d | Ixabepilone, 10 mg/d | Ixabepilone, 15 mg/d | Ixabepilone, 20 mg/d | Ixabepilone, 25 mg/d | Ixabepilone, 30 mg/d | Ixabepilone, MTD (25 mg), With Famotidine | Ixabepilone, MTD (25 mg), With Food
Started | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Ixabepilone With Famotidine or Food
Arm/Group | Ixabepilone, 5 mg/d | Ixabepilone, 10 mg/d | Ixabepilone, 15 mg/d | Ixabepilone, 20 mg/d | Ixabepilone, 25 mg/d | Ixabepilone, 30 mg/d | Ixabepilone, MTD (25 mg), With Famotidine | Ixabepilone, MTD (25 mg), With Food
Started | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ixabepilone, 5 mg/d: Participants with advanced cancer received daily oral doses of ixabepilone, 5 mg, on Days 1 through 5 every 21 days.
- Ixabepilone, 10 mg/d: Participants with advanced cancer received daily oral doses of ixabepilone, 10 mg, on Days 1 through 5 every 21 days.
- Ixabepilone, 15 mg/d: Participants with advanced cancer received daily oral doses of ixabepilone, 15 mg, on Days 1 through 5 every 21 days.
- Ixabepilone, 20 mg/d: Participants with advanced cancer received daily oral doses of ixabepilone, 20 mg, on Days 1 through 5 every 21 days.
- Ixabepilone, 25 mg/d: Participants with advanced cancer received daily oral doses of ixabepilone, 25 mg, on Days 1 through 5 every 21 days.
- Ixabepilone, 30 mg/d: Participants with advanced cancer received daily oral doses of ixabepilone, 30 mg, on Days 1 through 5 every 21 days.
- Total: Total of all reporting groups
Arm/Group | Ixabepilone, 5 mg/d | Ixabepilone, 10 mg/d | Ixabepilone, 15 mg/d | Ixabepilone, 20 mg/d | Ixabepilone, 25 mg/d | Ixabepilone, 30 mg/d | Total
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 23 | 6 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 2 | 2 | 21 | 3 | 32
  >=65 years | 2 | 3 | 1 | 1 | 2 | 3 | 12
Age, Continuous [Mean (Full Range); unit: years] | 64 [44 to 76] | 62 [43 to 72] | 60 [50 to 74] | 60 [49 to 73] | 56 [40 to 78] | 69 [63 to 83] | 60 [40 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 2 | 12 | 2 | 23
  Male | 1 | 3 | 1 | 1 | 11 | 4 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 2 | 0 | 4
  White | 3 | 5 | 2 | 3 | 17 | 6 | 36
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Death as Outcome, Treatment-related Adverse Events (AEs), and AEs Leading to Discontinuation
Description: An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition that does not necessarily have a causal relationship with treatment. Treatment related=possibly, probably, or certainly related to and of unknown relationship to study treatment.
Time Frame: Days 1 through 21 (Cycle 1), continuously
Population: All Treated Subjects: All subjects who received at least 1 dose of ixabepilone.
Measure: Number; unit: Participants
Groups:
- Ixabepilone, 5 mg/d: Participants received daily oral doses of ixabepilone, 5 mg, on Days 1-5 every 21 days. On all dosing days in Cycle 1, participants must fast at least 4 hours before and 4 hours after treatment. For Cycles 2 and greater, participants must fast 1 hour before and 2 hours after ixabepilone dose.
- Ixabepilone, 10 mg/d: Participants received daily oral doses of ixabepilone, 10 mg, on Days 1-5 every 21 days On all dosing days in Cycle 1, participants must fast at least 4 hours before and 4 hours after treatment. For Cycles 2 and greater, participants must fast 1 hour before and 2 hours after ixabepilone dose.
- Ixabepilone, 15 mg/d: Participants received daily oral doses of ixabepilone, 15 mg, on Days 1-5 every 21 days. On all dosing days in Cycle 1, participants must fast at least 4 hours before and 4 hours after treatment. For Cycles 2 and greater, participants must fast 1 hour before and 2 hours after ixabepilone dose.
- Ixabepilone, 20 mg/d: Participants received daily oral doses of ixabepilone, 20 mg, on Days 1-5 every 21 days. On all dosing days in Cycle 1, participants must fast at least 4 hours before and 4 hours after treatment. For Cycles 2 and greater, participants must fast 1 hour before and 2 hours after ixabepilone dose.
- Ixabepilone, 25 mg/d: Participants received daily oral doses of ixabepilone, 25 mg, on Days 1-5 every 21 days. On all dosing days in Cycle 1, participants must fast at least 4 hours before and 4 hours after treatment. For Cycles 2 and greater, participants must fast 1 hour before and 2 hours after ixabepilone dose.
- Ixabepilone, 30 mg/d: Participants received daily oral doses of ixabepilone, 30 mg, on Days 1-5 every 21 days. On all dosing days in Cycle 1, participants must fast at least 4 hours before and 4 hours after treatment. For Cycles 2 and greater, participants must fast 1 hour before and 2 hours after ixabepilone dose.
Arm/Group | Ixabepilone, 5 mg/d | Ixabepilone, 10 mg/d | Ixabepilone, 15 mg/d | Ixabepilone, 20 mg/d | Ixabepilone, 25 mg/d | Ixabepilone, 30 mg/d
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 23 | 6
Participants
  Death | 0 | 0 | 2 | 1 | 1 | 1
  Treatment-related AEs | 2 | 6 | 3 | 1 | 12 | 5
  AEs | 3 | 6 | 3 | 2 | 20 | 6
  AEs leading to discontinuation | 0 | 1 | 0 | 0 | 1 | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Ixabepilone
Description: MTD is based on Cycle 1 data only and defined as the maximum dose that can be administered to 6 participants with no more than 1 experiencing a dose-limiting toxicity (DLT) (or fewer than one third of participants if more than 6 receive treatment) with at least 2 participants experiencing a DLT at the next higher dose level. DLT=an event, such as neutropenia; thrombocytopenia; Gr 3 or 4 nausea or diarrhea; Gr 3 fatigue or asthenia; transient arthralgia or recalcitrant myalgia; and prolonged recovery from a toxicity, that occurs during the first course of treatment.
Time Frame: Days 1 through 21 (Cycle 1)
Population: All Treated Subjects: All subjects who received at least one dose of ixabepilone were included.
Measure: Number; unit: mg/d
Groups:
- All Treated Participants: Participants received daily oral doses of ixabepilone on Days 1-5 every 21 days. On all dosing days in Cycle 1, participants must fast at least 4 hours before and 4 hours after treatment. For Cycles 2 and greater, participants must fast 1 hour before and 2 hours after ixabepilone dose.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 44
mg/d | 25

3. Secondary Outcome: Number of Participants With Abnormal Laboratory Values by Worst CTC Grade
Description: Lower limit of normal (LLN)=lowest level of normal among all laboratory ranges. Hemoglobin (g/dL): Gr 1: 10.0-<LLN; Gr 2: 8.0-<10.0; Gr 3:6.5-<8.0; Gr 4: 6.5. Leukocytes (c/uL): Gr 1: 3.0-<LLN; Gr 2: 2.0-<3.0; Gr 3: 1.0-<2.0; Gr 4: <1.0. Lymphocytes (c/uL): Gr 1: 0.8-<1.5; Gr 2: 0.5-<0.8; Gr 3: 0.2-<0.5; Gr 4: <0.2. Neutrophils (Absolute)(c/uL): Gr 1: 1.5-<2.0; Gr 2: 1.0-<1.5; Gr 3: 0.5-<1.0; Gr 4: <0.5. Neutrophils + Bands (c/uL): Gr 1: 1.5-<2.0; Gr 2: 1.0-<1.5; Gr 3: 0.5-<1.0; Gr 4: <0.5. Platelet Count (c/uL):Gr 1: 75.0-<LLN; Gr 2: 50.0-<75.0; Gr 3: 25.0-<50.0; Gr 4: <25.0.
Time Frame: Baseline and Days 1, 8, and 15 of Cycle 1 (21 days)
Population: All Treated Subjects: All subjects who received at least one dose of ixabepilone were included.
Measure: Number; unit: Participants
Arm/Group | All Treated Participants
Number analyzed (Participants) | 44
Participants
  Hemoglobin (Grade 1) | 19
  Hemoglobin (Grade 2) | 15
  Hemoglobin (Grade 3) | 5
  Hemoglobin (Grade 4) | 0
  Leukocytes (Grade 1) | 7
  Leukocytes (Grade 2) | 4
  Leukocytes (Grade 3) | 2
  Leukocytes (Grade 4) | 3
  Lymphocytes (Absolute) (Grade 1) | 14
  Lymphocytes (Absolute) (Grade 2) | 14
  Lymphocytes (Absolute) (Grade 3) | 12
  Lymphocytes (Absolute) (Grade 4) | 3
  Neutrophils (Absolute) (Grade 1) | 3
  Neutrophils (Absolute) (Grade 2) | 0
  Neutrophils (Absolute) (Grade 3) | 1
  Neutrophils (Absolute) (Grade 4) | 4
  Neutrophils + Bands (Absolute) (Grade 1) | 3
  Neutrophils + Bands (Absolute) (Grade 2) | 0
  Neutrophils + Bands (Absolute) (Grade 3) | 1
  Neutrophils + Bands (Absolute) (Grade 4) | 4
  Platelet Count (Grade 1) | 3
  Platelet Count (Grade 2) | 3
  Platelet Count (Grade 3) | 1
  Platelet Count (Grade 4) | 1

4. Primary Outcome: Number of Participants With DLTs by Worst Common Terminology Criteria (CTC) Grade
Description: Adverse events (AEs) graded by CTC version 3. Grade (Gr) 1=mild; Gr 2=moderate; Gr 3=severe; Gr 4=life threatening; Gr 5=Death related to AE. DLT is defined as an event related to ixabepilone that occurs during the first course of treatment. Includes neutropenia; thrombocytopenia; Gr 3 or 4 nausea, vomiting, or diarrhea despite adequate medical intervention and prophylaxis; Gr 3 fatigue or asthenia; transient arthralgia or myalgia unresponsive to medical intervention; any Gr 3 nonhematologic toxicity; and prolonged recovery from a toxicity.
Time Frame: Days 1 through 21 (Cycle 1), continuously
Population: All Treated Participants: All participants who received at least one dose of ixabepilone were included.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 5 mg/d | Ixabepilone, 10 mg/d | Ixabepilone, 15 mg/d | Ixabepilone, 20 mg/d | Ixabepilone, 25 mg/d | Ixabepilone, 30 mg/d
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 23 | 6
Participants
  Clostridium difficile colitis (Grade 3) | 0 | 1 | 0 | 0 | 0 | 0
  Ileus (Grade 3) | 0 | 1 | 0 | 0 | 0 | 1
  Abdominal pain (Grade 3) | 0 | 0 | 0 | 0 | 0 | 1
  Fatigue (Grade 3) | 0 | 0 | 0 | 0 | 0 | 1
  Neutropenic fever (Grade 3) | 0 | 0 | 0 | 0 | 0 | 1
  Neutropenic fever (Grade 4) | 0 | 0 | 0 | 0 | 0 | 2
  Dehydration (Grade 3) | 0 | 0 | 0 | 0 | 0 | 1
  Diarrhea (Grade 3) | 0 | 0 | 0 | 0 | 0 | 2
  Hypokalemia (Grade 3) | 0 | 0 | 0 | 0 | 0 | 1
  Nausea (Grade 3) | 0 | 0 | 0 | 0 | 0 | 1
  Vomiting (Grade 3) | 0 | 0 | 0 | 0 | 0 | 1
  Mucosal inflammation (Grade 3) | 0 | 0 | 0 | 0 | 0 | 1
  Neutropenia (Grade 4) | 0 | 0 | 0 | 0 | 1 | 1
  Hypokalemia (Grade 4) | 0 | 0 | 0 | 0 | 1 | 0
  Hypophosphatemia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 1
  Thrombocytopenia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 1
  Sudden death (Grade 5) | 0 | 0 | 0 | 0 | 0 | 1

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Ixabepilone
Time Frame: Days 1 and 5 of Cycle 1
Population: All participants who received ixabepilone and who had adequate concentration profiles
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Ixabepilone, 5 mg/d; Ixabepilone, 10 mg/d; Ixabepilone, 15 mg/d; Ixabepilone, 20 mg/d; Ixabepilone, 25 mg/d; Ixabepilone, 30 mg/d: All participants who received ixabepilone and who had adequate concentration profiles were included.
Arm/Group | Ixabepilone, 5 mg/d | Ixabepilone, 10 mg/d | Ixabepilone, 15 mg/d | Ixabepilone, 20 mg/d | Ixabepilone, 25 mg/d | Ixabepilone, 30 mg/d
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 23 | 6
ng/mL
  Day1 (n=3, n=6, n=3, n=3, n=23, n=6) | 4.02 (1.99) | 25.93 (20.47) | 16.04 (16.76) | 24.10 (19.96) | 36.14 (25.18) | 43.67 (20.87)
  Day 5 (n=2, n=6, n=3, n=3, n=22, n=6) | 2.45 (0.42) | 20.34 (23.07) | 22.17 (12.40) | 32.73 (24.97) | 57.99 (99.77) | 66.48 (62.64)

6. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax) of Ixabepilone
Time Frame: Days 1 and 5 of Cycle 1
Population: All participants who received ixabepilone and who had adequate concentration profiles
Measure: Median (Full Range); unit: Hour
Arm/Group | Ixabepilone, 5 mg/d | Ixabepilone, 10 mg/d | Ixabepilone, 15 mg/d | Ixabepilone, 20 mg/d | Ixabepilone, 25 mg/d | Ixabepilone, 30 mg/d
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 23 | 6
Hour
  Day1 (n=3, n=6, n=3, n=3, n=23, n=6) | 2.0 [1.0 to 2.0] | 1.8 [1.0 to 3.0] | 4.0 [2.0 to 4.0] | 2.0 [2.0 to 3.0] | 2.0 [0.5 to 24.0] | 3.0 [1.5 to 4.0]
  Day 5 (n=2, n=6, n=3, n=3, n=22, n=6) | 2.3 [1.5 to 3.0] | 2.5 [1.0 to 5.0] | 5.0 [1.5 to 6.0] | 1.5 [1.5 to 2.0] | 1.8 [0.5 to 6.0] | 3.5 [2.0 to 8.0]

7. Secondary Outcome: Area Under the Concentration-time Curve in 1 Dosing Interval (AUC[TAU])of Ixabepilone
Time Frame: Days 1 and 5 of Cycle 1
Population: All participants who received ixabepilone and who had adequate concentration profiles.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Ixabepilone, 5 mg/d | Ixabepilone, 10 mg/d | Ixabepilone, 15 mg/d | Ixabepilone, 20 mg/d | Ixabepilone, 25 mg/d | Ixabepilone, 30 mg/d
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 23 | 6
ng*h/mL
  Day 1 (n=3, n=6, n=3, n=3, n=23, n=6) | 28.40 (29.73) | 91.79 (62.45) | 120.58 (152.23) | 120.82 (73.62) | 195.96 (177.39) | 252.01 (153.26)
  Day 5 (n=2, n=6, n=3, n=3, n=22, n=6) | 21.83 (28.59) | 143.85 (134.15) | 179.82 (126.95) | 222.73 (136.49) | 348.07 (370.95) | 545.42 (441.93)

8. Secondary Outcome: Plasma Half-life (T-Half) of Ixabepilone
Time Frame: Day 5 of Cycle 1
Population: All participants who received ixabepilone and who had adequate concentration profiles
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Ixabepilone, 5 mg/d | Ixabepilone, 10 mg/d | Ixabepilone, 15 mg/d | Ixabepilone, 20 mg/d | Ixabepilone, 25 mg/d | Ixabepilone, 30 mg/d
Number analyzed (Participants) | 2 | 6 | 3 | 3 | 22 | 6
Hours | 18.56 (NA) — Only 2 participants in this Arm on Day 5, so SD is not appropriate. | 47.00 (82.68) | 24.32 (17.68) | 35.25 (20.63) | 35.62 (17.48) | 34.14 (14.16)

9. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Oral Ixabepilone at MTD in Fasted and Fed Participants in Crossover Cohorts
Description: After the MTD has been defined, participants who completed Cycle 1 (ixabepilone, 25 mg, given once daily orally on Days 1 through 5 of 21-day cycle, with participants fasting at least 4 hours before and 4 hours after treatment on all dosing days) then cross over to Cycle 2, during which they consume a standard lowfat meal starting 30 minutes prior to ixabepilone, 25 mg, administration on Day 1 of Cycle 2 only. Meal is consumed within a 30-minute period. Administration of the total oral dose should not exceed more than 10 minutes from start to finish.
Time Frame: Up to 24 hours postdose Day 1 of Cycle 1 (21 days) and Day 1 of Cycle 2 (21 days)
Population: All participants who received ixabepilone and who had adequate concentration profiles. Participants received MTD (25 mg) ixabepilone without famotidine (Cycle 1) and then were crossed over to a cycle in which they received MTD (25 mg) ixabepilone with famotidine (Cycle 2).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ixabepilone, 25 mg/d
Number analyzed (Participants) | 8
ng/mL
  Fasted (Cycle 1) | 38.11 (29.48)
  Fed (Cycle 2) | 44.76 (38.69)

10. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax)of Oral Ixabepilone at MTD in Fasted and Fed Participants in Crossover Cohorts
Description: After the ixabepilone MTD (25 mg) has been defined, participants who completed Cycle 1 (ixabepilone, 25 mg, given once daily orally on Days 1 through 5 of 21-day cycle, with participants fasting at least 4 hours before and 4 hours after treatment on all dosing days) then cross over to Cycle 2, during which they consume a standard lowfat meal starting 30 minutes prior to ixabepilone, 25 mg, administration on Day 1 of Cycle 2 only. Meal is consumed within a 30-minute period. Administration of the total oral dose should not exceed more than 10 minutes from start to finish.
Time Frame: Up to 24 hours postdose Day 1 of Cycle 1 (21 days) and Day 1 of Cycle 2 (21 days)
Population: All participants who received ixabepilone and who had adequate concentration profiles. Participants received MTD (25 mg).
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Ixabepilone, 25 mg/d
Number analyzed (Participants) | 8
ng/mL
  Fasted (Cycle 1) | 2.0 [0.5 to 5.0]
  Fed (Cycle 2) | 4.0 [2.0 to 6.0]

11. Secondary Outcome: Area Under the Curve in 1 Dosing Interval (AUC[TAU]) of Oral Ixabepilone at MTD in Fasted and Fed Participants in Crossover Cohorts
Description: as for outcome 10
Time Frame: Up to 24 hours postdose Day 1 of Cycle 1 (21 days) and Day 1 of Cycle 2 (21 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Ixabepilone, 25 mg/d
Number analyzed (Participants) | 8
ng*h/mL
  Fasted (Cycle 1) | 190.22 (128.14)
  Fed (Cycle 2) | 243.46 (99.91)

12. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Oral Ixabepilone With and Without Famotidine in Crossover Cohorts
Description: After the ixabepilone MTD (25 mg) has been defined, participants who completed Cycle 1 (ixabepilone, 25 mg, given once daily orally on Days 1 through 5 of 21-day cycle, with participants fasting at least 4 hours before and 4 hours after treatment on all dosing days) then cross over to Cycle 2, during which they receive famotidine, 40 mg. Prior to dosing on Day 1 of Cycle 2, famotidine administered in an oral dose 2 hours before ixabepilone 25-mg dose.
Time Frame: Up to 24 hours postdose Day 1 of Cycle 1 (21 days) and Day 1 of Cycle 2 (21 days)
Population: Participants who received ixabepilone, at the MTD of 25 mg, alone in Cycle 1 and had adequate concentration profiles. Participants then were crossed over to a cycle in which they received MTD (25 mg) ixabepilone with famotidine,40 mg, on Day 1 of Cycle 2.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ixabepilone, 25 mg/d
Number analyzed (Participants) | 7
ng/mL
  Without Famotidine (Cycle 1) | 36.91 (29.79)
  With Famotidine (Cycle 2) | 66.16 (63.91)

13. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax) of Oral Ixabepilone With and Without Famotidine in Crossover Cohorts
Description: as for outcome 12
Time Frame: Up to 24 hours postdose Day 1 of Cycle 1 (21 days) and Day 1 of Cycle 2 (21 days)
Population: as for outcome 12
Measure: Median (Full Range); unit: ng/mL
Groups:
- Ixabepilone, 25 mg/d: Participants received MTD (25 mg) ixabepilone without famotidine (Cycle 1) and then were crossed over to a cycle in which they received MTD (25 mg) ixabepilone (with famotidine (Cycle 2). On all dosing days in Cycle 1, participants must fast at least 4 hours before and 4 hours after ixabepilone treatment. For Cycles 2 and greater, participants must fast 1 hour before and 2 hours after the dose.
Arm/Group | Ixabepilone, 25 mg/d
Number analyzed (Participants) | 7
ng/mL
  Without Famotidine (Cycle 1) | 3.0 [1.0 to 24.0]
  With Famotidine (Cycle 2) | 4.0 [2.0 to 6.0]

14. Secondary Outcome: Area Under the Curve in 1 Dosing Interval (AUC[TAU]) of Oral Ixabepilone With and Without Famotidine in Crossover Cohorts
Description: After the ixabepilone MTD (25 mg) has been defined, participants who completed Cycle 1 (ixabepilone, 25 mg, given alone once daily orally on Days 1 through 5 of 21-day cycle, with participants fasting at least 4 hours before and 4 hours after treatment on all dosing days) then cross over to Cycle 2, during which they receive famotidine, 40 mg. Prior to dosing on Day 1 of Cycle 2, famotidine administered in an oral dose 2 hours before ixabepilone 25-mg dose.
Time Frame: Up to 24 hours postdose Day 1 of Cycle 1 (21 days) and Day 1 of Cycle 2 (21 days)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Ixabepilone, 25 mg/d: Participants who received MTD (25 mg) ixabepilone without famotidine and then were crossed over to a cycle in which they received MTD (25 mg) ixabepilone with famotidine. Fasted/Fed criteria: Cycle 1: Dose 1 administered after a minimum of a 4-hour fast. Cycle 2: Dose 1 administered with a low-fat meal to crossover cohort.
Arm/Group | Ixabepilone, 25 mg/d
Number analyzed (Participants) | 7
ng*h/mL
  Without Famotidine (Cycle 1) | 218.36 (260.55)
  With Famotidine (Cycle 2) | 276.30 (179.20)

15. Secondary Outcome: Number of Participants With Significant Findings on Physical Examination or Electrocardiogram (ECG)
Description: Physical examination evaluated height, weight, Eastern Cooperative Oncology Group performance status, adverse events, and abnormal laboratory findings and included a neurologic examination to evaluate deep tendon reflexes, sensory modalities, and motor strength. Participants also underwent a 12-lead ECG screening. Physical examination findings and ECG findings were considered clinically significant at the investigator's discretion.
Time Frame: At screening and predose Day 1, Cycle 1 (21 days)
Population: Although physical examinations and ECGs were performed, the findings were not summarized.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 5 mg/d | Ixabepilone, 10 mg/d | Ixabepilone, 15 mg/d | Ixabepilone, 20 mg/d | Ixabepilone, 25 mg/d | Ixabepilone, 30 mg/d
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 23 | 6
Participants
  With abnormal physical examination findings | 0 | 0 | 0 | 0 | 0 | 0
  With abnormal ECG results | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Abnormal (CTC Grade 3 or Greater) Serum Chemistry Levels
Description: Upper limit of normal (ULN)=upper level of normal among all laboratory ranges. Alkaline phosphatase(U/L): Gr 3: >5.0-20.0*ULN; Gr 4: >20.0*ULN. Sodium (mEq/L): Gr 3: 120-<130 or >155-160; Gr 4 <120. Potassium (mEq/L): Gr 3: 2.5-<3.0 or >6.0-7.0; Gr 4: <2.5 or >7.0. Calcium (mg/dL): Gr 3: 6.0-<7.0 or >12.5-13.5; Gr 4: <6.0 or >13.5. Inorganic phosphorus (mg/dL): Gr 3: 1.0-<2.0; Gr 4: <1.0. Albumin (g/dL): Gr 3: <2.0.
Time Frame: At screening and predose Day 1, Cycle 1 (21 days)
Population: All Treated Subjects: All subjects who received at least one dose of ixabepilone were included.
Measure: Number; unit: Participants
Arm/Group | All Treated Participants
Number analyzed (Participants) | 44
Participants
  Low sodium (Grade 3) | 4
  High sodium (Grade 3) | 1
  Low albumin (Grade 3) | 3
  Low alkaline phosphatase (Grade 3) | 1
  Low potassium (Grade 3) | 1
  Low potassium (Grade 4) | 1
  Low total calcium (Grade 4) | 1
  Low inorganic phosphorus (Grade 4) | 1

ADVERSE EVENTS:
Groups:
- Ixabepilone, 5 mg: Participants received daily oral doses of ixabepilone, 5 mg, on Days 1-5 every 21 days
- Ixabepilone, 10 mg: Participants received daily oral doses of ixabepilone, 10 mg, on Days 1-5 every 21 days
- Ixabepilone, 15 mg: Participants received daily oral doses of ixabepilone, 15 mg, on Days 1-5 every 21 days
- Ixabepilone, 20 mg: Participants received daily oral doses of ixabepilone, 20 mg, on Days 1-5 every 21 days
- Ixabepilone, 25 mg: Participants received daily oral doses of ixabepilone, 25 mg, on Days 1-5 every 21 days
- Ixabepilone, 30 mg: Participants received daily oral doses of ixabepilone, 30 mg, on Days 1-5 every 21 days
Arm/Group | Ixabepilone, 5 mg | Ixabepilone, 10 mg | Ixabepilone, 15 mg | Ixabepilone, 20 mg | Ixabepilone, 25 mg | Ixabepilone, 30 mg
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/6 | 3/3 | 1/3 | 6/23 | 5/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 3/3 | 2/3 | 20/23 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone, 5 mg (N=3) | Ixabepilone, 10 mg (N=6) | Ixabepilone, 15 mg (N=3) | Ixabepilone, 20 mg (N=3) | Ixabepilone, 25 mg (N=23) | Ixabepilone, 30 mg (N=6)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 2 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Catheter-related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Noncardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Nonsmall cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone, 5 mg (N=3) | Ixabepilone, 10 mg (N=6) | Ixabepilone, 15 mg (N=3) | Ixabepilone, 20 mg (N=3) | Ixabepilone, 25 mg (N=23) | Ixabepilone, 30 mg (N=6)
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Culture urine positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Aphonia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 7 | 4
Vomiting (Gastrointestinal disorders) | 1 | 1 | 3 | 1 | 6 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 4 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 4 | 2
Abdominal mass (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastroesophogeal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Oncyhomyocosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 8 | 2
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 5 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 4 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 0 | 5 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 4 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 3 | 1
Chills (General disorders) | 1 | 1 | 0 | 0 | 3 | 2
Edema (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 4 | 1 | 1 | 13 | 3
Pyrexia (General disorders) | 0 | 4 | 1 | 0 | 3 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Implant site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Edema peripheral (General disorders) | 1 | 2 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
Noncardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acrohordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period <or=60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.